CLINICAL TRIAL: NCT04774393
Title: Phase 1b/2 Study of Oral Decitabine/Cedazuridine (ASTX727) and Venetoclax in Combination With the Targeted Mutant IDH1 Inhibitor Ivosidenib or the Targeted Mutant IDH2 Inhibitor Enasidenib
Brief Title: Decitabine/Cedazuridine and Venetoclax in Combination With Ivosidenib or Enasidenib for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1220; NCI-2021-00893 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1220 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; enasidenib; ivosidenib; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (decitabine/cedazuridine, venetoclax, ivosidenib) (Experimental): Patients receive decitabine/cedazuridine PO daily on days 1-5, venetoclax PO daily on days 1-14, and ivosidenib PO daily on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Ivosidenib; Drug: Venetoclax
- Arm B (decitabine/cedazuridine, venetoclax, enasidenib) (Experimental): Patients receive decitabine/cedazuridine PO daily on days 1-5, venetoclax PO daily on days 1-14, and enasidenib PO daily on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Enasidenib; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; Inqovi
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007 Free Base
  Arms: Arm B (decitabine/cedazuridine, venetoclax, enasidenib)
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
  Arms: Arm A (decitabine/cedazuridine, venetoclax, ivosidenib)
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trials studies the side effects of decitabine/cedazuridine (ASTX727) and venetoclax in combination with ivosidenib or enasidenib, and how well they work in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). ASTX727 is the combination of a fixed dose of 2 drugs, cedazuridine and decitabine. Cedazuridine may slow down how fast decitabine is broken down by the body, and decitabine may block abnormal cells or cancer cells from growing. Venetoclax may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Enasidenib and ivosidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving decitabine/cedazuridine and venetoclax in combination with ivosidenib or enasidenib may help control acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability and recommended phase 2 dose (RP2D) of oral decitabine/cedazuridine (ASTX727) and venetoclax in combination with either ivosidenib (Arm A) or enasidenib (Arm B) for patients with acute myeloid leukemia. (Phase Ib) II. To determine the overall response rate (complete response [CR], complete remission with incomplete hematologic recovery [CRh], morphologic leukemia-free state [MLFS] and partial response [PR)] of oral decitabine/cedazuridine (ASTX727) and venetoclax in combination with either ivosidenib (Arm A) or enasidenib (Arm B) for patients with acute myeloid leukemia. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine duration of response (DOR), event-free survival (EFS), and overall survival (OS).

II.To evaluate occurrence of minimal residual disease (MRD) negative status by multiparameter flow cytometry and molecular evaluation.

III. To determine the overall response rate (CR, CRh, Cri, MLFS and PR)

IV. Characterize the pharmacokinetic (PK) profiles of venetoclax in plasma samples (Phase 1b only)

EXPLORATORY OBJECTIVE:

I. To investigate global gene expression profiles, deoxyribonucleic acid (DNA) methylation profiles, BH3 profiling and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients receive decitabine/cedazuridine orally (PO) daily on days 1-5, venetoclax PO daily on days 1-14, and ivosidenib PO daily on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive decitabine/cedazuridine PO daily on days 1-5, venetoclax PO daily on days 1-14, and enasidenib PO daily on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of relapsed or refractory acute myeloid leukemia (AML) (including biphenotypic or bilineage leukemia including a myeloid component or isolated extramedullary AML); OR
* Patients (> 60 year old) with newly diagnosed AML not eligible for intensive chemotherapy are also eligible
* To be considered not eligible for intensive chemotherapy, participants must be defined by the following: Age 75 years or older, or Age 18 to 74 years with at least one of the following comorbidities:
* Severe cardiac disorder (eg, congestive heart failure requiring treatment, ejection fraction ≤50%, or chronic stable angina).
* Severe pulmonary disorder (eg, DLCO ≤65% or forced expiratory volume in 1 second [FEV1] ≤65%).
* Creatinine clearance ≥30 mL/min to <45 mL/min.
* Moderate hepatic impairment with total bilirubin >1.5 to ≤3.0 × upper limit of normal (ULN)
* ECOG performance status of 2 or 3
* Age >= 18 years
* Subjects must have documented IDH1 or IDH2 gene mutation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Adequate renal function including creatinine < 2 unless related to the disease
* Direct bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5 x ULN will be considered eligible)
* In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy agent(s). Oral hydroxyurea and/or cytarabine (up to 2 g/m^2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the principle investigator (PI). Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Male subjects who are sexually active with a women of childbearing potential (WOCBP) and who have not had vasectomies must be willing to use a barrier method of contraception and refrain from sperm donation from initial study drug until 90 days after last dose of study drug
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Patients with any concurrent uncontrolled clinically significant medical condition including life-threatening severe infection, or psychiatric illness, which could place the patient at unacceptable risk of study treatment
* Patients with active graft-versus-host-disease (GVHD) status post stem cell transplant (patients without active GVHD on chronic suppressive immunosuppression and/or phototherapy for chronic skin GVHD are permitted after discussion with the PI)
* Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications
* Corrected QT (QTc) interval using Fridericia's formula (QTcF) >= 450 msec. Bundle branch block and prolonged QTc interval are permitted after discussion with the PI
* Known active hepatitis B (HBV) or hepatitis C (HCV) infection or known human immunodeficiency virus (HIV) infection
* Subject has a white blood cell count > 25 x 10^9/L. (Note: Hydroxyurea is permitted to meet this criterion)
* Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception

  * Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double barrier methods (for example a condom in combination with a spermicide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (Phase Ib) | Up to 1 cycle (1 cycle = 28 days)
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5 by organ system.
Overall response rate (ORR) (Phase II) | Within 4 months of treatment
  Defined as complete remission (CR), CR with incomplete hematologic recovery, CR with incomplete count recovery, partial response or marrow clearance of blasts. Will estimate the ORR for the combination treatmen1t, along with the Bayesian 95% credible interval.
Incidence of adverse events (Phase II) | Within 4 months of treatment
  Assessed using Common Toxicity Criteria version 5.0. Safety data will be summarized using frequency and percentage, by category and severity.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Time interval between treatment start until disease progression, relapse/refractory, or death due to any cause, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of EFS. Log-rank tests will be used to compare among subgroups of patients in terms of EFS.
Overall survival (OS) | Time interval between treatment start until death due to any cause, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of OS. Log-rank tests will be used to compare among subgroups of patients in terms of OS.
Duration of response | Up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities and log-rank tests will be used to compare among subgroups of patients.
Minimal residual disease negative status | Up to 3 years
  Will be summarized graphically and with descriptive statistics. The association between molecular and cellular markers and overall response and/or resistance will be assessed through logistic regression analyses. Paired t-test or Wilcoxon signed rank test will be used to assess the marker change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] DiNardo CD, Marvin-Peek J, Loghavi S, Takahashi K, Issa GC, Jen WY, Daver NG, Reville PK, Short NJ, Sasaki K, Mullin JK, Bradley CA, Borthakur G, Maiti A, Alvarado Y, Pemmaraju N, Abbas HA, Hammond DE, Haddad F, Bravo GM, Chien KS, Yilmaz M, Kornblau SM, Jabbour E, Ravandi F, Kadia T, Garcia-Manero G, Konopleva MY, Kantarjian HM. Outcomes of Frontline Triplet Regimens With a Hypomethylating Agent, Venetoclax, and Isocitrate Dehydrogenase Inhibitor for Intensive Chemotherapy-Ineligible Patients With Isocitrate Dehydrogenase-Mutated AML. J Clin Oncol. 2025 Aug 20;43(24):2692-2699. doi: 10.1200/JCO-25-00640. Epub 2025 Jun 13. PMID 40513054
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04774393/ICF_000.pdf